CLINICAL TRIAL: NCT02150525
Title: A Randomized Trial to Explore the Effect of Oral Omega 3 Fatty Acids on Atrophic Vaginitis in Postmenopausal Breast Cancer Survivors
Brief Title: Effect of Omega 3 on Atrophic Vaginitis in Breast Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OSU-09145; NCI-2013-00068 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-08-19; First posted 2014-05-30 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Ductal Breast Carcinoma in Situ; Breast Cancer, Stage I; Breast Cancer, Stage II; Breast Cancer, Stage III
Keywords: breast cancer; vaginal dryness; dyspareunia; genital irritation
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms; Dyspareunia | interventions — Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (oral omega-3 fatty acid) (Experimental): Patients received 3.5g oral omega-3 fatty acid daily for 6 months. Questionnaire administration, pills counts, and medication diaries were collected at monthly intervals.
  Interventions: Dietary Supplement: omega-3 fatty acid; Behavioral: Questionnaire administration
- Arm II (placebo) (Placebo Comparator): Patients received equivalent, matched oral placebo (seven capsules) daily for 6 months. Questionnaire administration, pills counts, and medication diaries were collected at monthly intervals.
  Interventions: Other: placebo; Behavioral: Questionnaire administration

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acid — Given PO (by mouth) daily
  Other Names: fish oil; n-3 fatty acid; O3FA; PUFAs
  Arms: Arm I (oral omega-3 fatty acid)
Other: placebo — Given PO(by mouth)daily
  Other Names: PLCB
  Arms: Arm II (placebo)
Behavioral: Questionnaire administration — Measures of self-reported outcomes: Self-reported symptoms will be documented with the Urogenital Atrophy Questionnaire (UAQ), Menopausal Rating Scale (MRS), Female Sexual Function Index (FSFI), Center for Epidemiological Studies Short Depression Scale (CES-D 10), and Brief Pain Inventory (BPI).

SUMMARY:
This randomized double-blind clinical trial studied the effect of oral omega-3 fatty acid on atrophic vaginitis in postmenopausal breast cancer survivors (N=52). Omega-3 fatty acid may reduce inflammation and improve vaginal symptoms in postmenopausal breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the ability of oral omega-3 fatty acids to improve symptoms of atrophic vaginitis as reported by postmenopausal breast cancer survivors as compared to survivors not taking omega 3.

II.To examine the ability of oral omega-3 fatty acids to decrease inflammation related to atrophic vaginitis in postmenopausal breast cancer survivors as compared to survivors not taking omega 3.

III. To examine the ability of oral omega-3 fatty acids to uptake systemically and to validate adherence; these measures will be compared to demographic data including body mass index to observe if differences exist in postmenopausal breast cancer survivors vs. those not taking omega 3.

IV. To examine the effect of oral omega 3 fatty acids as compared to placebo of dietary supplement on serum female hormone levels in postmenopausal breast cancer survivors.

V. To examine cytokine levels in women taking oral omega 3 fatty acids as compared to women not taking omega 3 to determine effect.

OUTLINE: Patients were randomized to 1 of 2 treatment arms.

ARM I: Patients received 3.5g omega-3 fatty acid orally (PO) daily for 6 months.

ARM II: Patients received placebo of dietary supplement (7 capsules) PO daily for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Woman with a history of breast cancer, stage 0, I, II, or III
* At least 12 months from definitive surgical procedure (i.e. lumpectomy or mastectomy)
* At least 3 months from completion of chemotherapy
* Postmenopausal, defined as no menstrual cycle for 12 consecutive months, or surgical menopause
* Have one or more stated symptoms of atrophic vaginitis, such as vaginal dryness, genital irritation/itching, genital pain, and/or dyspareunia
* No current use of estrogen replacement therapy
* If recent use of estrogen replacement therapy, off at least three months
* No current use of estradiol-releasing vaginal ring or estradiol vaginal tablets; if recent use of these products, off at least 3 consecutive months
* No evidence of disease (NED), any cancer other than breast cancer
* No current use of oral omega 3 fatty acids or Vitamin E; if recent consistent use of these products, off at least six months; if sporadic use of these products, off at least 3 consecutive months
* May be taking oral anti-estrogens or aromatase inhibitors, and/or biologic therapy
* Must be willing to undergo venipuncture at 0, 3, and 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* No history of a bleeding tendency
* No history of uncontrolled hypertension, heart disease or stroke
* Hemoglobin > 10 g/dL
* Hematocrit > 30%
* White blood count > 3.5 K/uL
* Platelet count > 100,000/mm^3
* Fasting serum glucose < 115 mg/dL
* Total bilirubin < 1.6 mg/dL
* Transaminases alanine aminotransferase(ALT)and aspartate aminotransferase (AST)< 1.5 x ULN (upper limit of normal)

Exclusion Criteria:

* Metastatic malignancy of any kind
* Ongoing chemotherapy or radiation therapy (ongoing hormonal therapy and/or biologic therapy are allowed)
* History of pelvic or genital radiation therapy
* Use of Coumadin or other anticoagulants
* Known, active pelvic, vaginal, or urinary tract infections
* Current use of hormone replacement therapy, either systemic or local
* Uncontrolled co-morbidities including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable hypertension
* Psychiatric illness/social situation that would limit adherence to study requirements
* Consistent use of omega-3 fatty acid concentrates or capsules within the 6 months prior to entry on the study
* Known sensitivity or allergy to fish oil or omega 3 fish products
* Pregnant or nursing women
* Subjects who cannot give an informed consent

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Explore the ability of oral omega 3 fatty acids to improve symptoms of atrophic vaginitis as self-reported by postmenopausal breast cancer survivors that took omega 3 vs. those survivors who did not take omega 3. | From baseline to 3 and 6 months
  Self-reported measures included the Urogenital Atrophy Questionnaire, Brief Pain Inventory, Menopause Rating Scale, and Female Sexual Function Index. These measures were compared in women assigned to omega 3 fatty acids vs. women assigned to placebo of dietary supplement.

SECONDARY OUTCOMES:
Explore the ability of oral omega 3 fatty acids to decrease inflammation related to atrophic vaginitis in postmenopausal breast cancer survivors who took omega 3 fatty acids as compared to those survivors who did not take omega 3. | From baseline to 3 and 6 months
  This was measured by self-reported pain to touch during gynecological examination, self-reported vaginal dryness, pain, or irritation, wet prep results (presence or absence of yeast), pH, and parabasal layer that indicated a shift to less inflamed tissue, and gynecologic examination results.
Determine level of omega 3 uptake in those who took omega 3 vs. those who took placebo of dietary supplement by using tested serum levels of omega 3 fatty acids in all participants. | From baseline to 3 and 6 months
  Tested serum levels to evaluate the level of omega 3 fatty acids in women assigned to omega 3 vs. women assigned to placebo of dietary supplement to validate adherence and systemic uptake as compared to self-reported adherence and dietary records.
Measure if effects exist from omega 3 fatty acids by using tested serum hormone levels in all participants. | From baseline to 3 and 6 months
  The investigators tested serum hormone levels in women assigned to omega 3 fatty acids vs. women assigned to placebo of dietary supplement to determine the effect, if any, of omega 3 fatty acids.
Determine if an effect existed in women that took omega 3 fatty acids by using tested cytokine levels in all participants. | From baseline to 3 and 6 months
  Cytokine levels in women taking oral omega 3 fatty acids were tested and compared to cytokine levels in women not taking oral omega 3 fatty acids as compared to those women who did not take omega 3 fatty acids..

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Lester, PhD, CRNP, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Comprehensive Breast Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu